CLINICAL TRIAL: NCT05399290
Title: A Randomized Controlled Trial Investigating the Pediatric Patient Experience of Subantimicrobial Dose Doxycycline for Acne Treatment
Brief Title: Subantimicrobial Doxycycline in Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Michelle Gallagher, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003269
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Acne Vulgaris; Pediatrics
Keywords: Acne Vulgaris; Doxycycline; Sub-Antimicrobial; Pediatrics
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg standard dose doxycycline BID (Active Comparator): Oral, 12 weeks
  Interventions: Drug: Doxycycline Hyclate
- 20 mg sub-antimicrobial dose doxycycline BID (Experimental): Oral, 12 weeks
  Interventions: Drug: Doxycycline Hyclate

INTERVENTIONS:
Drug: Doxycycline Hyclate — 100 mg vs 20 mg doxycycline hyclate BID for 12 weeks

SUMMARY:
Antibiotic resistance is a public health problem that worsens the more physicians prescribe standard dose antibiotics for acne. Regardless of race, acne vulgaris is one of the most common dermatologic conditions among pediatric populations. As such, clinicians can make a large impact by practicing good antibiotic stewardship while still addressing the impact of acne on adolescents' self-esteem. Subantimicrobial doxycycline maintains its anti-inflammatory effects while eliminating antimicrobial properties and associated risks of drug resistance. Few studies, focused primarily on adults, have shown that subantimicrobial doxycycline is efficacious in treating acne from a physician standpoint. The investigators aim to investigate the patient experience of acne treatment with subantimicrobial dose doxycycline in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Documented moderate to severe facial acne

Exclusion Criteria:

* Other skin conditions on the face
* Previous antibiotic treatment for acne
* Use of antibiotics for any reason within the past month
* Use of new prescription regiment for acne within the last 3 months
* Positive pregnancy test in the clinic
* Cognitive impairments

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gallagher, DO, Principal Investigator — Michigan State University
Locations (1):
- Messenger Dermatology Clinic, Lansing, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 100 mg Standard Dose Doxycycline BID | 20 mg Sub-antimicrobial Dose Doxycycline BID
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg Standard Dose Doxycycline BID | 20 mg Sub-antimicrobial Dose Doxycycline BID | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Patient Perceptions of Their Acne Treatment
Description: Biweekly Qualtrics surveys were administered to identify changes in the self-reported severity of facial acne lesions using a 10-point ordinal Likert-type scale at 7 post-prescription time point (week 0, week 2, week 4, week 6, week 8, week 10, week 12). The minimum value is 1 and the maximum value is 10, with increasing acne severity (i.e. 10 is most severe acne).
  * In the table below, participants are labelled by a letter (A, B, etc.) to differentiate the different time points (rows) but participants in each treatment group (100 mg vs 20 mg) are different and not related.
  * Data is missing for timepoints when surveys were not submitted
Time Frame: 12 weeks
Population: 10 participants in each group were analyzed as they had fulfilled the requirement of submitting a minimum of 3 survey ratings out of 7 total (week 0, 2, 4, 6, 8, 10, 12). A total of 62 ratings were analyzed in the 100 mg treatment arm (i.e. there were 8 surveys not submitted among the 10 participants), and 56 ratings in the 20 mg treatment arm.
Measure: Number; unit: score on a scale
Units Other Than Participants: Survey Ratings
Arm/Group | 100 mg Standard Dose Doxycycline BID | 20 mg Sub-antimicrobial Dose Doxycycline BID
Number analyzed (Participants) | 10 | 10
Number analyzed (Survey Ratings) | 62 | 56
score on a scale
  Week 0 (A): number analyzed (Participants) | 1 | 1
  Week 0 (A): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (A) | 8 | 8
  Week 2 (A): number analyzed (Participants) | 1 | 1
  Week 2 (A): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (A) | 7 | 7
  Week 4 (A): number analyzed (Participants) | 1 | 1
  Week 4 (A): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (A) | 8 | 7
  Week 6 (A): number analyzed (Participants) | 1 | 1
  Week 6 (A): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (A) | 9 | 6
  Week 8 (A): number analyzed (Participants) | 1 | 1
  Week 8 (A): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (A) | 8 | 7
  Week 10 (A): number analyzed (Participants) | 0 | 1
  Week 10 (A): number analyzed (Survey Ratings) | 0 | 1
  Week 10 (A) |  | 4
  Week 12 (A): number analyzed (Participants) | 0 | 1
  Week 12 (A): number analyzed (Survey Ratings) | 0 | 1
  Week 12 (A) |  | 4
  Week 0 (B): number analyzed (Participants) | 1 | 1
  Week 0 (B): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (B) | 8 | 6
  Week 2 (B): number analyzed (Participants) | 1 | 1
  Week 2 (B): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (B) | 8 | 7
  Week 4 (B): number analyzed (Participants) | 1 | 1
  Week 4 (B): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (B) | 6 | 6
  Week 6 (B): number analyzed (Participants) | 1 | 1
  Week 6 (B): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (B) | 5 | 5
  Week 8 (B): number analyzed (Participants) | 1 | 1
  Week 8 (B): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (B) | 5 | 6
  Week 10 (B): number analyzed (Participants) | 1 | 0
  Week 10 (B): number analyzed (Survey Ratings) | 1 | 0
  Week 10 (B) | 3 |
  Week 12 (B): number analyzed (Participants) | 1 | 0
  Week 12 (B): number analyzed (Survey Ratings) | 1 | 0
  Week 12 (B) | 2 |
  Week 0 (C): number analyzed (Participants) | 1 | 1
  Week 0 (C): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (C) | 7 | 6
  Week 2 (C): number analyzed (Participants) | 1 | 1
  Week 2 (C): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (C) | 6 | 6
  Week 4 (C): number analyzed (Participants) | 1 | 0
  Week 4 (C): number analyzed (Survey Ratings) | 1 | 0
  Week 4 (C) | 5 |
  Week 6 (C): number analyzed (Participants) | 1 | 1
  Week 6 (C): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (C) | 3 | 4
  Week 8 (C): number analyzed (Participants) | 1 | 1
  Week 8 (C): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (C) | 3 | 4
  Week 10 (C): number analyzed (Participants) | 1 | 1
  Week 10 (C): number analyzed (Survey Ratings) | 1 | 1
  Week 10 (C) | 3 | 3
  Week 12 (C): number analyzed (Participants) | 0 | 1
  Week 12 (C): number analyzed (Survey Ratings) | 0 | 1
  Week 12 (C) |  | 4
  Week 0 (D): number analyzed (Participants) | 1 | 1
  Week 0 (D): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (D) | 8 | 7
  Week 2 (D): number analyzed (Participants) | 1 | 1
  Week 2 (D): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (D) | 8 | 7
  Week 4 (D): number analyzed (Participants) | 1 | 1
  Week 4 (D): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (D) | 8 | 8
  Week 6 (D): number analyzed (Participants) | 1 | 0
  Week 6 (D): number analyzed (Survey Ratings) | 1 | 0
  Week 6 (D) | 7 |
  Week 8 (D): number analyzed (Participants) | 1 | 0
  Week 8 (D): number analyzed (Survey Ratings) | 1 | 0
  Week 8 (D) | 7 |
  Week 10 (D): number analyzed (Participants) | 0 | 0
  Week 10 (D): number analyzed (Survey Ratings) | 0 | 0
  Week 12 (D): number analyzed (Participants) | 1 | 0
  Week 12 (D): number analyzed (Survey Ratings) | 1 | 0
  Week 12 (D) | 6 |
  Week 0 (E): number analyzed (Participants) | 1 | 1
  Week 0 (E): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (E) | 8 | 6
  Week 2 (E): number analyzed (Participants) | 1 | 1
  Week 2 (E): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (E) | 6 | 6
  Week 4 (E): number analyzed (Participants) | 1 | 0
  Week 4 (E): number analyzed (Survey Ratings) | 1 | 0
  Week 4 (E) | 4 |
  Week 6 (E): number analyzed (Participants) | 1 | 1
  Week 6 (E): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (E) | 0 | 6
  Week 8 (E): number analyzed (Participants) | 1 | 1
  Week 8 (E): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (E) | 8 | 5
  Week 10 (E): number analyzed (Participants) | 0 | 1
  Week 10 (E): number analyzed (Survey Ratings) | 0 | 1
  Week 10 (E) |  | 5
  Week 12 (E): number analyzed (Participants) | 0 | 1
  Week 12 (E): number analyzed (Survey Ratings) | 0 | 1
  Week 12 (E) |  | 5
  Week 0 (F): number analyzed (Participants) | 1 | 1
  Week 0 (F): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (F) | 6 | 7
  Week 2 (F): number analyzed (Participants) | 1 | 0
  Week 2 (F): number analyzed (Survey Ratings) | 1 | 0
  Week 2 (F) | 5 |
  Week 4 (F): number analyzed (Participants) | 1 | 1
  Week 4 (F): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (F) | 5 | 7
  Week 6 (F): number analyzed (Participants) | 1 | 1
  Week 6 (F): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (F) | 5 | 6
  Week 8 (F): number analyzed (Participants) | 1 | 1
  Week 8 (F): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (F) | 5 | 7
  Week 10 (F): number analyzed (Participants) | 1 | 1
  Week 10 (F): number analyzed (Survey Ratings) | 1 | 1
  Week 10 (F) | 4 | 4
  Week 12 (F): number analyzed (Participants) | 1 | 0
  Week 12 (F): number analyzed (Survey Ratings) | 1 | 0
  Week 12 (F) | 5 |
  Week 0 (G): number analyzed (Participants) | 1 | 1
  Week 0 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (G) | 5 | 6
  Week 2 (G): number analyzed (Participants) | 1 | 1
  Week 2 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (G) | 3 | 6
  Week 4 (G): number analyzed (Participants) | 1 | 1
  Week 4 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (G) | 3 | 6
  Week 6 (G): number analyzed (Participants) | 1 | 1
  Week 6 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (G) | 4 | 7
  Week 8 (G): number analyzed (Participants) | 1 | 1
  Week 8 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (G) | 5 | 7
  Week 10 (G): number analyzed (Participants) | 1 | 1
  Week 10 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 10 (G) | 3 | 6
  Week 12 (G): number analyzed (Participants) | 1 | 1
  Week 12 (G): number analyzed (Survey Ratings) | 1 | 1
  Week 12 (G) | 2 | 5
  Week 0 (H): number analyzed (Participants) | 1 | 1
  Week 0 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (H) | 8 | 7
  Week 2 (H): number analyzed (Participants) | 1 | 1
  Week 2 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (H) | 7 | 6
  Week 4 (H): number analyzed (Participants) | 1 | 1
  Week 4 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (H) | 8 | 5
  Week 6 (H): number analyzed (Participants) | 1 | 1
  Week 6 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (H) | 7 | 4
  Week 8 (H): number analyzed (Participants) | 1 | 1
  Week 8 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (H) | 7 | 3
  Week 10 (H): number analyzed (Participants) | 1 | 1
  Week 10 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 10 (H) | 6 | 2
  Week 12 (H): number analyzed (Participants) | 1 | 1
  Week 12 (H): number analyzed (Survey Ratings) | 1 | 1
  Week 12 (H) | 7 | 2
  Week 0 (I): number analyzed (Participants) | 0 | 1
  Week 0 (I): number analyzed (Survey Ratings) | 0 | 1
  Week 0 (I) |  | 6
  Week 2 (I): number analyzed (Participants) | 1 | 1
  Week 2 (I): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (I) | 5 | 4
  Week 4 (I): number analyzed (Participants) | 1 | 1
  Week 4 (I): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (I) | 3 | 6
  Week 6 (I): number analyzed (Participants) | 1 | 1
  Week 6 (I): number analyzed (Survey Ratings) | 1 | 1
  Week 6 (I) | 3 | 4
  Week 8 (I): number analyzed (Participants) | 1 | 1
  Week 8 (I): number analyzed (Survey Ratings) | 1 | 1
  Week 8 (I) | 2 | 5
  Week 10 (I): number analyzed (Participants) | 1 | 1
  Week 10 (I): number analyzed (Survey Ratings) | 1 | 1
  Week 10 (I) | 2 | 4
  Week 12 (I): number analyzed (Participants) | 1 | 1
  Week 12 (I): number analyzed (Survey Ratings) | 1 | 1
  Week 12 (I) | 2 | 3
  Week 0 (J): number analyzed (Participants) | 1 | 1
  Week 0 (J): number analyzed (Survey Ratings) | 1 | 1
  Week 0 (J) | 8 | 9
  Week 2 (J): number analyzed (Participants) | 1 | 1
  Week 2 (J): number analyzed (Survey Ratings) | 1 | 1
  Week 2 (J) | 7 | 10
  Week 4 (J): number analyzed (Participants) | 1 | 1
  Week 4 (J): number analyzed (Survey Ratings) | 1 | 1
  Week 4 (J) | 6 | 8
  Week 6 (J): number analyzed (Participants) | 1 | 0
  Week 6 (J): number analyzed (Survey Ratings) | 1 | 0
  Week 6 (J) | 7 |
  Week 8 (J): number analyzed (Participants) | 1 | 0
  Week 8 (J): number analyzed (Survey Ratings) | 1 | 0
  Week 8 (J) | 6 |
  Week 10 (J): number analyzed (Participants) | 0 | 0
  Week 10 (J): number analyzed (Survey Ratings) | 0 | 0
  Week 12 (J): number analyzed (Participants) | 1 | 0
  Week 12 (J): number analyzed (Survey Ratings) | 1 | 0
  Week 12 (J) | 5 |
Statistical Analysis 1: Comparison: 100 mg Standard Dose Doxycycline BID vs 20 mg Sub-antimicrobial Dose Doxycycline BID; Test type: Other — Chi square analysis was conducted to detect any significant between group differences (100 mg vs 20 mg) in perceived acne severity; p = 0.677, Chi-squared
Statistical Analysis 2: Comparison: 100 mg Standard Dose Doxycycline BID; Test type: Other — Friedman's test was conducted for the 100 mg treatment arm to detect any significant within group differences in perceived acne severity; p = 0.002, Friedman's test
Statistical Analysis 3: Comparison: 20 mg Sub-antimicrobial Dose Doxycycline BID; Test type: Other — Friedman's test was conducted for the 20 mg treatment arm to detect any significant within group differences in perceived acne severity; p = 0.018, Fried

2. Other Pre Specified Outcome: Changes in Medication, Open Comments in the Qualtrics Survey Regarding Acne Treatment
Description: Participants are invited to report any medication changes and submit open-ended comments concerning their use of doxycycline or their acne experiences.
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Side Effects
Description: Any side effects associated with taking doxycycline for acne is encouraged to be discussed with the clinician
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | 100 mg Standard Dose Doxycycline BID | 20 mg Sub-antimicrobial Dose Doxycycline BID
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Standard Dose Doxycycline BID (N=11) | 20 mg Sub-antimicrobial Dose Doxycycline BID (N=11)
Photoallergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
No Improvement (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT05399290/Prot_SAP_ICF_000.pdf